CLINICAL TRIAL: NCT01902758
Title: Enhancing Physical Performance and Mitigating Acute Mountain Sickness Via Pharmaceutical Intervention While at Altitude
Brief Title: Drug Combination on Exercise Performance at High Altitude
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Montana (Other)
Responsible Party: Principal Investigator, Brent Ruby, Director of the Montana Center for Work Physiology and Exercise Metabolism, University of Montana
Allocation: Non-Randomized | Model: Parallel | Masking: Triple
Other Study IDs: UM82-13; N66001-10-C-2134 (Other Grant/Funding Number: DARPA)
Record Dates: First submitted 2013-07-11; First posted 2013-07-18 (Estimated); Results first posted 2016-01-25 (Estimated); Last update posted 2016-02-26 (Estimated); Status verified 2016-01

CONDITIONS: Acute Mountain Sickness
Keywords: exercise performance
MeSH Terms: conditions — Altitude Sickness | interventions — ambrisentan; Theophylline

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- ambrisentan and theophylline (Experimental): ambrisentan (5mg) once daily for 2 consecutive days theophylline (400mg) once daily for 2 consecutive days
  Interventions: Drug: ambrisentan and theophylline
- placebo (Placebo Comparator): matched placebo tablets wil be given at the same time to the comparison group as the medications to the experimental group
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: ambrisentan and theophylline
  Arms: ambrisentan and theophylline
Drug: placebo — placebo for comparison group
  Arms: placebo

SUMMARY:
This study is being conducted to determine the effectiveness of using two FDA approved medications in concert to reduce the likelihood of sickness due to low oxygen levels and to reduce the decrement in physical performance at higher elevations. The investigators hypothesize that this drug combination will reduce the symptoms of acute mountain sickness and improve exercise performance at high altitude compared to placebo.

ELIGIBILITY:
Inclusion Criteria:

* healthy males

Exclusion Criteria:

* VO2max below 45ml/kg/min
* currently taking any medication

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2013-08; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Montana Center for Work Physiology and Exercise Metabolism, Missoula, Montana, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Ambrisentan and Theophylline: ambrisentan (5mg) once daily for 2 consecutive days theophylline (400mg) once daily for 2 consecutive days
  ambrisentan and theophylline
Period: Overall Study
Arm/Group | Ambrisentan and Theophylline | Placebo
Started | 14 | 14
Completed | 14 | 14
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ambrisentan and Theophylline | Placebo | Total
Number analyzed (Participants) | 14 | 14 | 28
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 14 | 14 | 28
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 22 (2) | 23 (2) | 23 (2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 14 | 14 | 28
Region of Enrollment [Number; unit: participants]
  United States | 14 | 14 | 28

OUTCOME MEASURES:

1. Primary Outcome: Time (Minutes) to Complete 2 Miles on a Treadmill
Time Frame: after arriving at high altitude (within 1 hour)
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Ambrisentan and Theophylline | Placebo
Number analyzed (Participants) | 14 | 14
seconds | 1544 (109) | 1540 (158)

ADVERSE EVENTS:
Arm/Group | Ambrisentan and Theophylline | Placebo
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/14
Other Adverse Events (participants affected / at risk) | 0/14 | 0/14

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No